CLINICAL TRIAL: NCT03471884
Title: Effects of Nonintubated Thoracoscopic Lobectomy on Lung Protection: A Randomized Controlled Trial
Brief Title: Effects of Nonintubated Thoracoscopic Lobectomy on Lung Protection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201711003RINB
Record Dates: First submitted 2018-03-13; First posted 2018-03-21 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Non-small Cell Lung Cancer; Lung Function Decreased; Tracheal Intubation Morbidity
Keywords: Thoracoscopic surgery,Airway Management,Anesthesia
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nonintubated thoracoscopic lobectomy (Experimental): Lung cancer patients undergoing thoracoscopic lobectomy without tracheal intubation
  Interventions: Procedure: Nonintubated thoracoscopic lobectomy
- Intubated thoracoscopic lobectomy (Active Comparator): Lung cancer patients undergoing thoracoscopic lobectomy with tracheal intubation and one-lung ventilation
  Interventions: Procedure: Intubated thoracoscopic lobectomy

INTERVENTIONS:
Procedure: Nonintubated thoracoscopic lobectomy — Nonintubated general anesthesia using fentanyl, target-controlled infusion of propofol to achieve a bispectral index value between 40 and 60. One-lung ventilation will be achieved via a spontaneous breathing due to iatrogenic pneumothorax.
  Arms: Nonintubated thoracoscopic lobectomy
Procedure: Intubated thoracoscopic lobectomy — Intubated general anesthesia using 2%-3% sevoflurane and rocuronium to achieve a bispectral index value between 40 and 60. One-lung ventilation will be achieved via a endobronchial tube or blocker with use of mechanical ventilation.
  Arms: Intubated thoracoscopic lobectomy

SUMMARY:
A novel nonintubated thoracoscopic technique is promising to enhance recovery after thoracic surgery. However, the effects of nonintubated technique on specific organ protection in not clear yet. In this randomized trial, the effect of nonintubated technique on lung function protection will be evaluated via PaO2/FiO2 ratio, oxidative stress and inflammatory cytokines serially in lung cancer patients undergoing thoracoscopic lobectomy.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related death worldwide. Its incidence is increasingly arising recently. For early-stage non-small cell lung cancer, surgery is the standard treatment that offers best chance of survival. For thoracoscopic lung cancer surgery, tracheal intubation with one-lung ventilation is regarded the standard anesthetic management to establish a safe operating environment. However, complications associated with intubated general anesthesia are not negligible. A novel nonintubated thoracoscopic technique is developing and applied in a variety of thoracic diseases. A previous study showed that nonintubated thoracoscopic lobectomy was feasible and safe in lung cancer patients. Furthermore, nonintubated techniques was also associated with a faster recovery of oral intake, less postoperative complications and shorter hospital stay. The effects of nonintubated thoracoscopic technique on specific organ protection is not clear yet.

The aim of this investigation is to explore the effects of nonintubated thoracoscopic lobectomy on lung function protection in lung cancer patients, comparing with the standard intubated patients as a control. The investigators are going to enrol 82 lung cancer patients and randomize them equally to complete thoracoscopic lobectomy with lymphadenectomy either with a nonintubated technique (n=41) or an intubated technique (n=41). The assessment of lung function will be obtained from serial blood gas analyses using PaO2/FiO2 ratio. Additionally, oxidative stress and inflammatory cytokines will be measured from serial blood samples including 8-isoprostane, malondialdehyde, tumor necrosis factor-α, interleukin-6, interleukin-10, S100-β and neuron specific enolase.

ELIGIBILITY:
Inclusion criteria

* adults (> 20 year-old), lung cancer patients undergoing thoracoscopic lobectomy

Exclusion criteria

* obesity (BMI > 26 kg/m2)
* previous ipsilateral thoracic surgery
* severe ventilatory insufficiency (oxygen/BiPAP user)
* poor cardiopulmonary function (preop forced expiratory volume at one second (FEV1) <60%, preop left ventricular ejection fraction < 50%)
* autoimmune disease requiring chronic steroids
* patients with difficult airway management, pregnant women

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Lung function assessment | 12 hours
  Lung function will be assessed by serial arterial blood gas analyses to obtain oxygenation index (PaO2/FiO2).

SECONDARY OUTCOMES:
Oxidative and systemic inflammatory cytokines. | 24 hours
  Oxidative and systemic inflammatory cytokines will be measured from serial blood samples, including 8-isoprostane (pg/mL), malondialdehyde (nM), tumor necrosis factor-alpha (pg/mL), interleukin-6 (pg/mL), interleukin-10 (pg/mL), S100-beta (pg/mL), and neuron specific enolase (ng/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Hui Hung, MD, MSc, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan